CLINICAL TRIAL: NCT03186222
Title: Polymorphism of Extrapituitary Promoter of PRL Gene and Relationships With Serum Prolactin Levels in Acne Vulgaris.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Mostafa Tawfik, principal investigator, Assiut University
Other Study IDs: POEPOPRGAGARWSPLIAV
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases with acne vulgaris: A group of 100 patients with acne vulgaris. blood sample are taken in the morning hours, between 08:00 and 10:00 am.
  Interventions: Diagnostic Test: blood sample
- control group: control group of 100 age and sex matched healthy volunteers. blood sample are taken in the morning hours, between 08:00 and 10:00 am.
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — Serum PRL levels are measured using ELISA assay kit in both groups and correlated with severity of acne in acne group.
  The genomic DNA from peripheral leukocytes is extracted. Genotyping of 1149G/T single nucleotide polymorphism (SNP) PRL extrapituitary promoter is done in acne patients and healthy individuals (control group) using PCR-RFLP method.

SUMMARY:
Acne vulgaris is one of the most common skin diseases. It is a disease of the pilosebaceous units, clinically characterized by seborrhea, comedones, papules, pustules, nodules and, in some cases, scarring.

DETAILED DESCRIPTION:
The pathogenesis of acne has been attributed to multiple factors such as increased sebum production, alteration of the quality of sebum lipids, regulation of cutaneous steroidogenesis, androgen activity, interaction with neuropeptides, exhibition of pro- and anti- inflammatory properties, follicular hyperkeratinization and the action of Propionibacterium acnes (P. acnes) within the follicle .

Central or peripheral stress may induce the development of clinical inflammation in the pilosebaceous unit, leading to the development of acne lesions or to exacerbation of pre-existing acne . Prolactin is one of the major hormonal signals that are immediately upregulated on psychoemotional and physical stress .

The discovery of locally produced extrapituitary prolactin and that human skin is both a source and target of prolactin production has increased interest in cutaneous prolactin research . Prolactin and prolactin receptors expression have now been demonstrated in several cutaneous cell populations, including keratinocytes, fibroblasts, sweat glands and sebaceous glands. Hence, prolactin is likely to be involved as a mediator in the ''brain-skin axis'' .

Given that the mammary gland is an epidermal derivative, it is not surprising that the pilosebaceous unit, another epidermal derivative, has also surfaced as a prominent, non-classical prolactin target organ expressing prolactin receptors .

In human skin, Prolactin and prolactin receptors are both expressed in the sebaceous gland , and prolactin stimulates sebum production . These effects are evident in women with hyperprolactinemia, who develop hirsutism and seborrhea, not uncommonly associated with female pattern balding . Patients treated with hyperprolactinemia-inducing neuroleptic agents also develop seborrhea . As sebocytes are prominent target cells of neuroendocrine signaling , prolactin might also contribute to the aggravating effect of psychoemotional stress on acne vulgaris. Besides the stimulation of sebocyte proliferation, which enhances holocrine secretion of this gland, this might also be related to effects on peripheral androgen metabolism .

The secretion of extrapituitary prolactin is regulated by the alternative promoter of prolactin gene , and the G/T polymorphism in position -1149 seems to be associated with level of prolactin expression .

In view of the recognized increase of human prolactin serum levels upon psychoemotional stress and the exacerbating effect of psychological stress on acne, together with a proposed role of prolactin in acne pathogenesis, it would be interesting to investigate the role of prolactin in acne vulgaris

ELIGIBILITY:
Inclusion Criteria: patients with acne vulgaris.

Exclusion Criteria:

* patients below 12 years of age
* patients recieving disorders and drug that could alter levels of prolactin such as thyroid disorders, renal and/or hepatic failure and drug use.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A group of 100 patients with acne vulgaris and another control group of 100 age and sex matched healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
polymorphism of extrapituitary promoter of PRL gene in acne cases and controls | 1 year
  The blood samples are taken in the morning hours, between 08:00 and 10:00 am The genomic DNA from peripheral leukocytes is extracted. Genotyping of 1149G/T single nucleotide polymorphism (SNP) PRL extrapituitary promoter is done in acne patients and healthy individuals (control group) using PCR-RFLP method.
  The genomic DNA from peripheral leukocytes is extracted. Genotyping of 1149G/T single nucleotide polymorphism (SNP) PRL extrapituitary promoter is done in acne patients and healthy individuals (control group) using PCR-RFLP method.

SECONDARY OUTCOMES:
serum prolactin levels in acne patients and controls and among different acne severity grades | 1 year
  The blood samples are taken in the morning hours, between 08:00 and 10:00 am. Serum PRL levels are measured using ELISA assay kit in both groups and correlated with severity of acne in acne group.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Awad, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zouboulis CC, Eady A, Philpott M, Goldsmith LA, Orfanos C, Cunliffe WC, Rosenfield R. What is the pathogenesis of acne? Exp Dermatol. 2005 Feb;14(2):143-52. doi: 10.1111/j.0906-6705.2005.0285a.x. PMID 15679586
- [Background] Ganceviciene R, Graziene V, Bohm M, Zouboulis CC. Increased in situ expression of melanocortin-1 receptor in sebaceous glands of lesional skin of patients with acne vulgaris. Exp Dermatol. 2007 Jul;16(7):547-52. doi: 10.1111/j.1600-0625.2007.00565.x. PMID 17576233
- [Background] Arck PC, Slominski A, Theoharides TC, Peters EM, Paus R. Neuroimmunology of stress: skin takes center stage. J Invest Dermatol. 2006 Aug;126(8):1697-704. doi: 10.1038/sj.jid.5700104. PMID 16845409
- [Background] Oakes SR, Rogers RL, Naylor MJ, Ormandy CJ. Prolactin regulation of mammary gland development. J Mammary Gland Biol Neoplasia. 2008 Mar;13(1):13-28. doi: 10.1007/s10911-008-9069-5. Epub 2008 Jan 25. PMID 18219564
- [Background] Zouboulis CC, Schagen S, Alestas T. The sebocyte culture: a model to study the pathophysiology of the sebaceous gland in sebostasis, seborrhoea and acne. Arch Dermatol Res. 2008 Sep;300(8):397-413. doi: 10.1007/s00403-008-0879-5. Epub 2008 Aug 9. PMID 18690467
- [Background] Langan EA, Ramot Y, Goffin V, Griffiths CE, Foitzik K, Paus R. Mind the (gender) gap: does prolactin exert gender and/or site-specific effects on the human hair follicle? J Invest Dermatol. 2010 Mar;130(3):886-91. doi: 10.1038/jid.2009.340. Epub 2009 Nov 5. No abstract available. PMID 19890346
- [Background] Reem GH, Ray DW, Davis JR. The human prolactin gene upstream promoter is regulated in lymphoid cells by activators of T-cells and by cAMP. J Mol Endocrinol. 1999 Jun;22(3):285-92. doi: 10.1677/jme.0.0220285. PMID 10343287
- [Background] Paus R. Does prolactin play a role in skin biology and pathology? Med Hypotheses. 1991 Sep;36(1):33-42. doi: 10.1016/0306-9877(91)90161-q. PMID 1766412